CLINICAL TRIAL: NCT01903668
Title: Determination of the Nature of the Endogenous Ligand of TREM-1 and Its Use as a New Diagnostic Biomarker in Sepsis
Status: Withdrawn | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Ducoroy PHRC IR 2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Step 1: Identification and characterisation of the TREM1L protein from samples already available characterised at the hospital Central of Nancy Step 2: Study of the isoforms of TREM1L in correlation with the prognosis of sepsis, Step 3: implementation of assay methods for TREM1L (ELISA or SUPRA MS) Step 4: Validation of assays for TREM1L and its isoforms in a larger number of subjects (inclusion of samples from Dijon CHU and Besançon CHU)

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalised in a Medical Intensive Care unit whatever the reason
* written informed consent obtained

Exclusion Criteria:

* patients less than 18 years old or under guardianship, persons without national health insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood samples used for this study come from a collection being created as part of the research entitled "The combined determination STREM-1/PCT/CD64 it allows the diagnosis of sepsis in intensive care" - No. IDRCB 2009 - A00870-57 and led by Professor Sebastian GIBOT CHU Nancy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
plasma concentrations of sTREM-1 | baseline